CLINICAL TRIAL: NCT03728543
Title: Efficacy and Safety Study of Sugammadex in Children 0-2 Years Old
Brief Title: the Efficacy and Safety of Sugammadex in Children 0-2 Years Old
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2018-04
Record Dates: First submitted 2018-06-25; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Anesthesia; Pediatric Cancer; Pediatric Tumor; Pediatric Hepatoblastoma; Beta-Thalassemia; Hepatic Metastases
Keywords: Anesthesia; Pediatrics; Pediatric oncology; MRI anesthesia
MeSH Terms: conditions — Neoplasms; Hepatoblastoma; beta-Thalassemia | interventions — Sugammadex

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children 0-2yo (Experimental): Children 0-2 years old with oncological diseases who need an MRI under general anesthesia, will receive sugammadex 2mg/kg IV
  Interventions: Drug: Sugammadex
- Children 2-18yo (Active Comparator): Children 2-18 years old with oncological diseases who need an MRI under general anesthesia, will receive sugammadex 2mg/kg IV
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — Introductory anesthesia: sevoflurane up to 8 rev /% + Air + O2 or propofol 1% 2 mg / kg intravenously.
  Maintenance: sevoflurane up to 3 rev /% + Air + O2, introduction of rocuronium bromide in a dose of 0.4 mg / kg, intravenously, as a bolus injection.
  At the end of anesthesia: sugammadex in a dose of 2 mg / kg, intravenously, as a bolus injection
  Other Names: Bridion

SUMMARY:
Sugammadex is a selective antidote to muscle relaxants rocuronium bromide and vecuronium bromide. Sugammadex is a modified gamma-cyclodextrin, a compound that selectively binds rocuronium bromide and vecuronium bromide. It forms a complex with them in the blood plasma, which leads to the decrease in the concentration of muscle relaxant binding to nicotinic receptors in the neuromuscular synapse. The result is the the elimination of neuromuscular blockade caused by rocuronium bromide or vecuronium bromide. Sugammadex is used to eliminate neuromuscular blockade caused by rocuronium bromide in children aged 2 years and adolescents in standard clinical situations. The aim of the study is to prove the efficacy and safety of sugammadex in children under 2 years

DETAILED DESCRIPTION:
Nowadays muscle relaxants are widely used in pediatric practice, but their use is fraught with numerous risks and complications. The main ones are the residual neuromuscular block and the possibility of developing a recurrence in the patient. In connection with this, the development and introduction into practical anesthesiology of new, more effective drugs for arresting the action of muscle relaxants is still relevant.

One of the them, sugammadex was recently introduced into clinical practice and provided a fundamentally new approach to the recovery of neuromuscular conduction. Often, children under two years of age need general anesthesia for MRI (prolonged stay in the device, apnea to get a high-quality image without respiratory artifacts, severe pain syndrome, severe neurological deficit, etc.). The aim of the study is the evaluation of the efficacy of sugammadex, estimated by restoring neuromuscular conduction within 0-120 seconds after bolus administration, and the safety and tolerability of sugammadex in children under two years of age. Children will be observed in the hospital during 24 hours. A group of patients from 2 to 18 years of age, in whom the drug sugammadex is used as standard therapy will be taken as a comparison group .

ELIGIBILITY:
Inclusion Criteria:

* Children 0 to 2 years (0 - 24 months, inclusive) in the study group; children from 2 to 18 years in the comparison group (control group)
* Patients with malignant neoplasms of the liver, malignant neoplasms with metastatic liver damage, beta-thalassemia
* Informed consent of the patient and / or parents or trustee of the patient

Exclusion Criteria:

* kidney failure
* liver failure
* critical conditions
* septicemia
* severe and decompensated diseases of the cardiovascular system
* refusal of the patient and / or his parents or trustee to participate in the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-11-20 (Estimated)

PRIMARY OUTCOMES:
Recovery time of neuromuscular conduction | 2 minutes post dose
  The time of the elimination of neuromuscular blockade (in seconds)

SECONDARY OUTCOMES:
Toxicity | 90 minutes after the injection
  Assessment of all adverse events from the time of injection to the time of leaving of the MRI department
Long-term toxicity | 24 hours post-dose
  Assessment of all adverse events during next 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anna Konstantinova, MD, Principal Investigator — Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 month of study completionData
Access Criteria: data access requests will be reviewed by the chief investigator and the local administration